CLINICAL TRIAL: NCT03508245
Title: Investigating Circadian Rhythms in Youth With Persistent Tic Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Emily J. Ricketts, PhD, Principal Investigator, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-000869; K23MH113884-01 (NIH)
Record Dates: First submitted 2018-04-16; First posted 2018-04-25 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Tourette's Disorder
Keywords: Tourette Syndrome; Tourette's; Tics; Circadian; Sleep
MeSH Terms: conditions — Tourette Syndrome; Tics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Wearable short wavelength light therapy (Other): Wearable short wavelength light therapy
  Interventions: Other: Wearable short wavelength light therapy

INTERVENTIONS:
Other: Wearable short wavelength light therapy — Wearable short wavelength (i.e., blue-green) light-emitting glasses worn for two weeks
  Other Names: Re-Timer

SUMMARY:
This study examines circadian rhythms and morningness-eveningness preference in youth with Persistent Tic Disorders (PTDs), including Tourette's Disorder (TD); and assesses the effects of wearable short wavelength light therapy on circadian rhythms and tic symptoms.

DETAILED DESCRIPTION:
Many individuals with Persistent Tic Disorders (PTDs), including Tourette's Disorder (TD) fail to significantly benefit from existing tic treatments. Case studies have shown morning exposure to light therapy, known to advance circadian phase is associated with modest to large tic reductions (Coles & Strauss, 2013; Niederhofer, 2003) suggesting the presence of circadian abnormalities (i.e., phase delay) in select individuals with PTDs. The present project assesses circadian phase and morningness-eveningness preference in youth with Persistent Tic Disorders (PTDs), including Tourette's Disorder (TD), and examines whether morning use of wearable short wavelength light therapy is associated with shifts in circadian rhythms and reductions in tic severity.

Study participation will take place over a three-week period. Clinician-rated tic interview and rating scales of morningness-eveningness preference, sleep, tic, and other symptoms will be completed during an initial screening assessment. Participants will then monitor sleep at home using an actigraph for one week and return for a baseline clinical assessment of tic severity and evening assessment of internal melatonin levels involving saliva sampling every 30 minutes for 6.5 hours in a dimly lit room. Next, participants will complete an abbreviated course (i.e., two weeks) of morning light therapy using wearable short wavelength (i.e., blue-green) light-emitting glasses while continuing to monitor sleep using the actigraph. Following this two-week period participants will return for a final assessment of tic severity and internal melatonin levels.

ELIGIBILITY:
Inclusion Criteria:

1. DSM-5 diagnosis of Tourette's Disorder, Persistent Motor Tic Disorder, or Persistent Vocal Tic Disorder
2. Yale Global Tic Severity Scale Score ≥ 14 for Tourette's Disorder or ≥ 10 for Persistent Motor Tic Disorder or Persistent Vocal Tic Disorder
3. fluency in English

Exclusion Criteria:

1. Current or lifetime diagnosis of Bipolar Disorder, psychosis, or autism spectrum disorder
2. Suicidality, severe depression or anxiety (i.e., Depression or anxiety diagnosis is more severe than Tourette's Disorder; equivalence in severity is allowed), or substance dependence, present within the past 6 months
3. Current diagnosis of Obstructive Sleep Apnea, Restless leg syndrome, Periodic Limb Movement Disorder, or Narcolepsy
4. Intellectual functioning below the low average range (WASI-II IQ score < 80)
5. Hypnotic medications, or melatonin within 8 weeks of study enrollment
6. Changes in dosage of any psychiatric medications within the past month
7. Behavior therapy for tics within the past 3 months
8. Prior use of light therapy
9. Current pregnancy or travel across > 2 time zones in the past month
10. Medical or neurological condition (e.g., seizure disorder, migraines) that would interfere in the individual's ability to participate in the study

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2018-01-18 (Actual); Primary Completion 2023-06-23 (Actual); Study Completion 2023-06-23 (Actual)

PRIMARY OUTCOMES:
Dim Light Melatonin Onset | 2 weeks
  The clock time at which salivary melatonin concentration reaches a threshold of 4 picograms (pg) per milliliter.
Yale Global Tic Severity Scale (YGTSS) | 2 weeks
  The YGTSS (Leckman et al., 1989) is a clinician-administered measure of tic severity encompassing tic number, frequency, intensity, complexity, and interference. The measure yields independent severity ratings for motor and vocal tics, a combined total tic severity score (0 to 50), and an independent tic-related impairment score (0 to 50).

SECONDARY OUTCOMES:
Clinical Global Impression-Improvement (CGI-I) Scale | 2 weeks
  The CGI-I (Guy, 1976) is a clinician-rated scale that has been used in a number of clinical trials for over 25 years, and in several studies with TD patients. The CGI-I is a clinician-rated measure of global patient improvement relative to baseline based on the clinician's perspective. Scores of Much (2) or Very Much (1) Improved indicate positive treatment response.
Children's Morningness-Eveningness Preferences Scale (CMEP) | 2 weeks
  The CMEP (Carskadon et al., 1993) is a 10-item measure of diurnal or nocturnal activity preference in recent past weeks. It will be modified to assess symptoms in the past week for the present study. The measure yields a total score ranging from 10 (extreme evening preference) to 42 (extreme morning preference).
Parent Tic Questionnaire (PTQ) | 2 weeks
  The PTQ (Chang et al., 2008) is a parent-reported measure of tic severity assessing both motor and vocal tics present within the past week. Individual tics are rated separately according to frequency and intensity. The measure yields separate scores for motor and vocal tics, in addition to a combined total tic severity score.

CONTACTS AND LOCATIONS:
Overall Officials: Emily J Ricketts, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- Semel Institute for Neuroscience and Human Behavior, University of California, Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carskadon MA, Vieira C, Acebo C. Association between puberty and delayed phase preference. Sleep. 1993 Apr;16(3):258-62. doi: 10.1093/sleep/16.3.258. PMID 8506460
- [Background] Chang S, Himle MB, Tucker BTP, Woods DW. Initial psychometric properties of a brief-parent-report instrument for assessing tic severity in children with chronic tic disorders. Child and Family Behavior Therapy 31(3): 181-191, 2009.
- [Background] Coles ME, Strauss GP. Shedding light on tics. Psychiatry Res. 2015 Feb 28;225(3):743. doi: 10.1016/j.psychres.2014.12.024. Epub 2014 Dec 23. No abstract available. PMID 25571772
- [Background] Guy W. ECDEU assessment manual for psychopharmacology. Rev. Rockville, Md.: National Institute of Mental Health. (DHEW publication no. (ADM) 76-338), 1976.
- [Background] Leckman JF, Riddle MA, Hardin MT, Ort SI, Swartz KL, Stevenson J, Cohen DJ. The Yale Global Tic Severity Scale: initial testing of a clinician-rated scale of tic severity. J Am Acad Child Adolesc Psychiatry. 1989 Jul;28(4):566-73. doi: 10.1097/00004583-198907000-00015. PMID 2768151
- [Background] Niederhofer H. Bright light therapy may be a therapeutic option for Tourette's syndrome. Acta Neuropsychologica 7(4): 283-285, 2009.